CLINICAL TRIAL: NCT00396045
Title: A Multicenter, Open Label Study of Oral Melphalan, Prednisone, and CC-5013 (Revlimid) (MPR) as Induction Therapy in Elderly Newly Diagnosed Multiple Myeloma Patients
Brief Title: Melphalan, Prednisone, and CC-5013 (Revlimid) as Induction Therapy in Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-026; MPR
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma, Lenalidomide, elderly patients
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

INTERVENTIONS:
Drug: Revlimid (CC-5013)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the association of Melphalan/Prednisone/Revlimid (MPR) as induction treatment for newly diagnosed myeloma patients over age 65 or those under 65 years who refuse or are not eligible for high dose therapy. This association might further increase the response rate achieved by the standard oral MP regimen.

DETAILED DESCRIPTION:
In Multiple Myeloma patients, the standard treatment is the oral combination of Melphalan and Prednisone (MP). This approach induces a partial response (PR) rate of approximately 50% and a complete remission (CR) rate of 1-5%, with a median remission duration of 18-20 months and a median overall survival of 3 years.

Recently, the combination of oral MP plus thalidomide increased response rate to 80% and complete remission rate to 20%, marked cytoreduction is the first step toward a sustained remission period.

CC-5013 (Revlimid) is a thalidomide analogue, 50000 times more potent than thalidomide in inhibiting TNF-alfa secretion, a potent growth factor for myeloma cells. Revlimid represents a novel class of anti-cancer drugs, it is active in patients with multiple myeloma who are refractory to conventional and high-dose chemotherapy with a response rate of approximately 30%. The association Revlimid plus dexamethasone further increases the response rate induced by Revlimid by an additional 30%.

This study will evaluate the safety and efficacy of the association of Melphalan/Prednisone/Revlimid (MPR) as induction treatment for newly diagnosed myeloma patients over age 65 or those under 65 years who refuse or are not eligible for high dose therapy. This association might further increase the response rate achieved by the standard oral MP regimen.

In the first part of the study (phase I component), different doses of oral Melphalan (0.18-0.25 mg/Kg) associated with Prednisone (MP) will be combined with escalating doses of Revlimid (from 5 mg/day) and administered together. This phase will define the MTD of the association. In the second part of the study (phase II component), 30 patients will be treated with MPR at dose/s defined from phase I component to verify data of response and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of a legally consenting age as defined by local regulations.
* Age > 65 years or age < 65 years in patients who refuse or are not eligible for high-dose therapy.
* Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal for 24 consecutive months or surgically sterilised or agree to continuous abstinence from heterosexual sexual contact or willing to use two acceptable method of birth control at the same time (one highly effective method and one additional effective method)(Highly Effective Methods: Intrauterine device -IUD-; Hormonal -birth control pills, injections, implants-; tubal ligation; partner's vasectomy; Additional Effective Methods: Latex condom; Diaphragm; Cervical Cap) for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of Lenalomide therapy - Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of Lenalomide therapy.
* Patient was previously diagnosed with symptomatic multiple myeloma based on standard criteria, and has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours; measurable plasmacytoma as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan); bone marrow plasma cells >10%.
* Patient has a Karnofsky performance status ≥ 60%
* Patient has a life-expectancy > 6 months.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):
* Absolute neutrophil count > 1.5 x 109/L without the use of growth factors
* Platelet count > 75 x 109/L without transfusion support within 7 days before the test.
* Calculated or measured creatinine clearance: ≥ 20 mL/minute
* Total bilirubin < 1.5 x the ULN
* AST (SGOT) and ALT (SGPT) < 2.5 x ULN
* Corrected serum calcium ≤ 14 mg/dL (3.5 mmol/L

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or beast feeding females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other concomitant standard/experimental anti-myeloma drug or therapy.
* Any prior use of CC-5013 or other anti-myeloma therapy.
* Any of the following laboratory abnormalities:
* Platelet count < 75 x 109/L.
* Absolute neutrophil count <1.5 x 109/L.
* Calculated or measured creatinine clearance <20 mL/minute.
* Corrected serum calcium >14 mg/dL (3.5 mmol/L).
* Aspartate transaminase (AST): >2.5 x the upper limit of normal (ULN).
* Alanine transaminase (AST): > 2.5 x the ULN.
* Total bilirubin: > 1.5 x the ULN.
* Known positive for HIV or active infectious hepatitis, type B or C.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54
Dates: Start 2005-01; Study Completion 2008-01

PRIMARY OUTCOMES:
SAFETY AND EFFICACY

SECONDARY OUTCOMES:
PROGRESSION FREE SURVIVAL AND OVERALL SURVIVAL

CONTACTS AND LOCATIONS:
Overall Officials: MARIO BOCCADORO, MD, Principal Investigator — DIVISIONE DI EMATOLOGIA DELL'UNIVERSITA' DI TORINO, AZIENDA OSPEDALIERA SAN GIOVANNI BATTISTA, TORINO, ITALY; ANTONIO PALUMBO, MD, Study Director — DIVISIONE UNIVERSITARIA DI EMATOLOGIA, AZIENDA OSPEDALIERA SAN GIOVANNI BATTISTA, TORINO, ITALY
Locations (9):
- Italy (9):
  - Unità Operativa di Ematologia, Spedali Civili, Brescia, Brescia
  - Reparto di Ematologia, Ospedale Ferrarotto, Catania, Catania
  - Unità Operativa Complessa Di Ematologia, Presidio Ospedaliero Dell'Annunziata, Azienda Ospedaliera Di Cosenza, Cosenza, COSENZA
  - Unità Operativa di Ematologia Trapianto di Cellule Staminali, Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Clinica Ematologica, Ospedale San Martino -Università di Genova, Genova, Genova
  - Cattedra di Ematologia, Dipart. Di Medicina Interna e Scienze Biomediche, Parma, Parma
  - Divisione di Ematologia-Policlinico Umberto I-Università La Sapienza, Roma, Roma
  - Divisione di Ematologia, Azienda Ospedaliera Senese Ospedale A. Sclavo, Siena, Siena
  - Div. Univ. Di Ematologia, Az. Osp. San Giovanni Battista, Torino, TORINO

REFERENCES:
- [Background] Palumbo A, Bertola A, Musto P, Caravita T, Callea V, Nunzi M, Grasso M, Falco P, Cangialosi C, Boccadoro M. Oral melphalan, prednisone, and thalidomide for newly diagnosed patients with myeloma. Cancer. 2005 Oct 1;104(7):1428-33. doi: 10.1002/cncr.21342. PMID 16116606
- [Background] Dimopoulos MA, Anagnostopoulos A, Weber D. Treatment of plasma cell dyscrasias with thalidomide and its derivatives. J Clin Oncol. 2003 Dec 1;21(23):4444-54. doi: 10.1200/JCO.2003.07.200. PMID 14645435
- [Background] Richardson PG, Schlossman RL, Weller E, Hideshima T, Mitsiades C, Davies F, LeBlanc R, Catley LP, Doss D, Kelly K, McKenney M, Mechlowicz J, Freeman A, Deocampo R, Rich R, Ryoo JJ, Chauhan D, Balinski K, Zeldis J, Anderson KC. Immunomodulatory drug CC-5013 overcomes drug resistance and is well tolerated in patients with relapsed multiple myeloma. Blood. 2002 Nov 1;100(9):3063-7. doi: 10.1182/blood-2002-03-0996. PMID 12384400
- [Background] Kraut EH, Crowley JJ, Wade JL, Laufman LR, Alsina M, Taylor SA, Salmon SE. Evaluation of topotecan in resistant and relapsing multiple myeloma: a Southwest Oncology Group study. J Clin Oncol. 1998 Feb;16(2):589-92. doi: 10.1200/JCO.1998.16.2.589. PMID 9469346
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033